CLINICAL TRIAL: NCT06094998
Title: Health Status of Children Born After Assisted Reproductive Technologies With the Development of Prediction Model and Principles of Child Management.
Brief Title: Health Status of Children Born After Assisted Reproductive Technologies
Status: Completed | Type: Observational
Sponsor: Kazakhstan's Medical University "KSPH" (Other)
Collaborators: Vyacheslav Notanovich Lokshin (Unknown); Nurgalieva Zhanar Zhenisovna (Unknown); Manzhuova Lyazzat Nurbapayevna (Unknown); Abshekenova Aigerim Temirkhanovna (Unknown); Valeria Nekhorosheva (Unknown); Kusainova Farida Azimovna (Unknown)
Responsible Party: Principal Investigator, Sevara Ilmuratova, PhD candidate, Researcher, Kazakhstan's Medical University "KSPH"
Other Study IDs: ИРН AP14872103
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Children Born After Assisted Reproductive Technologies; Health Status; Child Development
Keywords: children born after assisted reproductive technologies; health status; in vitro fertilization; assisted reproductive technologies; infertility; children's health; morbidity patterns; endocrine status; immunological status; congenital malformations; maternal age; physical development
MeSH Terms: conditions — Infertility; Congenital Abnormalities | interventions — CD4 Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children born after ART: 120 children born after assisted reproductive technologies
  Interventions: Diagnostic Test: hemogram examination
- children conceived spontaneously: 132 children conceived spontaneously
  Interventions: Diagnostic Test: hemogram examination

INTERVENTIONS:
Diagnostic Test: hemogram examination — It will be studied hemogram examination, immunity indicators (cellular components CD3, CD4, CD8, CD16, CD20, CD25, CD95, CD3 HLA DR+, CD# HLA-DR; humoral components - IgM, IgA, IgE, IgG) and laboratory investigations in endocrine system (TSH, free T3 and T4 levels, insulin, insulin-like growth factor-1 (IGF-1), somatotropic hormone (STH); glucose, potassium, sodium) in 120 children born after ART. Researchers will compare 132 children conceived spontaneously to see if ART can influent on the health status in future.
  Other Names: immunity indicators (cellular components CD3, CD4, CD8, CD16, CD20, CD25, CD95, CD3 HLA DR+, CD# HLA-DR; humoral components - IgM, IgA, IgE, IgG); laboratory investigations in endocrine system (TSH, free T3 and T4 levels, insulin, insulin-like growth factor-1 (IGF-1), somatotropic hormone (STH); glucose, potassium, sodium)

SUMMARY:
The goal of this observational study is to study the features of psychophysical development and the morbidity patterns of children born after assisted pregnancy, and to identify the connection with the health status of mothers, followed by the development of a prediction model and general principles of management of children born after ART. The main questions it aims to answer are: • the influence of premorbid background of mothers on children's physical development, disease occurrence and morbidity patterns of children born as after ART.

* To identify the indicators of cellular and humoral immunity in children born after different oocyte fertilization methods in IVF programs (classical IVF or ICSI).
* To study the long-term effects of ART on the endocrine status of children.

It will be studied hemogram examination, immunity indicators (cellular components CD3, CD4, CD8, CD16, CD20, CD25, CD95, CD3 HLA DR+, CD# HLA-DR; humoral components - IgM, IgA, IgE, IgG) and laboratory investigations in endocrine system (TSH, free T3 and T4 levels, insulin, insulin-like growth factor-1 (IGF-1), somatotropic hormone (STH); glucose, potassium, sodium) in 120 children born after ART. Researchers will compare 132 children conceived spontaneously to see if ART can influent on the health status in future.

DETAILED DESCRIPTION:
The tasks of the planned scientific and engineering project are based on the study of health status of children born after ART. The presence of a large cohort of children after ART in Kazakhstan will allow us to study morbidity patterns with the connection of mother's anamnesis, as well as to develop a prediction model and algorithms for the management of children conceived by assisted pregnancy. A comprehensive assessment of the health status of children born after ART will make it possible to determine the effect of the method of conception on the risks of immunity-related diseases and endocrine system pathology. It will allow us to predict deviations and ensure timely access to specialists and further examination. The presence of a burdened psychological background in couples with infertility may further influence the psychosocial adaptation of children conceived by ART and/or provoke higher morbidity rates in this group of children. It is important for the healthy and full integration of these children into society, including successful professional development in the future.

2.2. The project objective: to study the features of psychophysical development and the morbidity patterns of children born after assisted pregnancy, and to identify the connection with the health status of mothers, followed by the development of a prediction model and general principles of management of children born after ART.

Project Tasks

1. To study the influence of premorbid background of mothers on children's physical development, disease occurrence and morbidity patterns of children based on a retrospective study of 120 medical records of mothers and their children born as after ART.
2. To determine the indicators of cellular and humoral immunity (hemogram examination, cellular components CD3, CD4, CD8, CD16, CD20, CD25, CD95, CD3 HLA DR+, CD# HLA-DR; humoral components - IgM, IgA, IgE, IgG) in children born after ART.
3. To study the long-term effects of the hormone therapy in 120 mothers on the endocrine status (TSH, free T3 and T4 levels, insulin, insulin-like growth factor-1 (IGF-1), somatotropic hormone (STH); glucose, potassium, sodium) of children born after ART.
4. To develop a prediction model and algorithms for the management of children born after ART.

ELIGIBILITY:
Inclusion Criteria:

* successful ART program after IVF and ICSI,
* the transfer of fresh and frozen-thawed embryos (FET)
* a single or multiple pregnancy
* the birth of a child in the period from 2017 to 2023.

Exclusion Criteria:

* intrauterine insemination
* ART programs with donor gametes
* surrogacy.

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: To determine the characteristics of the health status of children born after assisted reproductive technologies, a study was conducted on the basis of the Scientific Center of Pediatrics and Pediatric Surgery, the PERSONA International Clinical Center for Reproductology and the Institute of Reproductive Medicine in Almaty
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Immune status of children born after assisted reproductive technologies | 1 day over which each participant is assessed
  hemogram examination(leycosytes, lymphosytes), immunity indicators (cellular components CD3, CD4, CD8, CD16, CD20, CD25, CD95, CD3 HLA DR+, CD# HLA-DR; humoral components - IgM, IgA, IgE, IgG)
laboratory investigations in endocrine system | 1 day over which each participant is assessed
  TSH, free T3 and T4 levels, insulin, insulin-like growth factor-1 (IGF-1), somatotropic hormone (STH); glucose, potassium, sodium

SECONDARY OUTCOMES:
Anthropometric measures | 1 day over which each participant is assessed
  assessment of Weight-for-age (kg), Weight-for-length/height, assessment of Length/height-for-age (cm), assessment of Head circumference for age (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Sevara K Ilmuratova, Principal Investigator — Kazakhstan Medical University "KSPH"; Vyacheslav Lokshin, PhD, Study Chair — International Clinical Centre of Reproduction "PERSONA"; Lyazzat Manzhuova, PhD, Study Chair — Scientific Center of Pediatrics and Pediatric Surgery; Zhanar Nurgaliyeva, PhD, Principal Investigator — Asfendiyarov Kazakh National Medical University; Farida Kussainova, MD, Principal Investigator — Asfendiyarov Kazakh National Medical University; Аygul Bazarbaeva, MD, Study Director — Scientific Center of Pediatrics and Pediatric Surgery; Valeriya Nekhorosheva, MD, Principal Investigator — Institute of Reproductive Medicine; Aygerim Abshekenova, MD, Principal Investigator — International Clinical Centre of Reproduction "PERSONA"
Locations (1):
- Scientific Center of Pediatrics and Pediatric Surgery, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided